CLINICAL TRIAL: NCT06299202
Title: Contrast-enhanced Spectral Mammography (CESM) Early Quantitative Evaluation of Tumoral Response and Pathologic Complete Response Prediction for Localized Breast Cancer Treated by Neoadjuvant Chemotherapy
Acronym: CERePred
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL23_0204; ID-RCB (Other: 2023-A01905-40)
Record Dates: First submitted 2024-02-19; First posted 2024-03-07 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Contrast Enhanced Spectral Mamography; Neodjuvant chemotherapy; Quantitative analysis; Complete histological response
MeSH Terms: conditions — Breast Neoplasms | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with localized breast cancer (Experimental): Patients with localized breast cancer (stage II or III, HER 2, triple-negative) eligible for a neoadjuvant chemotherapy and not presenting contraindication to angiomammography.
  Interventions: Diagnostic Test: Diagnostic test

INTERVENTIONS:
Diagnostic Test: Diagnostic test — * Inclusion visit (V1) Initial baseline CESM (V2) 15 days after inclusion
  * First chemotherapy treatment (V3) 28 days after V2.
  * Unilateral follow-up CESM (V4) 4 to 6 weeks after the first course of chemotherapy.
  * Surgery (V5):
    3 to 6 weeks later at the end of the complete treatment with primary chemotherapy
  * End of research visit (V6) It corresponds to the histological analysis on the surgical specimen after the complete treatment with neoadjuvant or primary chemotherapy.

SUMMARY:
Some types of localised breast cancer, including stage II and III, HER2 positive (Human Epidermal Growth Factor Receptor) or triple negative cancers are treated with primary or neoadjuvant chemotherapy prior to surgical treatment (mastectomy or conservative treatment).

Follow-up with neoadjuvant or primary chemotherapy is usually done by breast Magnetic Resonance Imaging (MRI).Tumour response to treatment is assessed on morphological size criteria.

Angiomammography (also called CESM : Contrast Enhanced Spectral Mammography) is an innovative and validated imaging technique consisting of dual energy mammography with injection of iodinated contrast medium; two images are generated, one comparable to a standard mammography and a second image highlighting the structures enhanced by the contrast medium. The characteristic neo angiogenesis of the tumour process thus allows good visualisation of the tumour compared to the underlying mammary gland.

A classical morphological analysis is therefore possible thanks to standard mammographic acquisition coupled with a quantitative functional analysis linked to the study of enhancement.

During angiomammography, several images are acquired in succession, starting with the cranio caudal view and ending with the profile view. On the same examination, these acquisitions are carried out at different injection times, making it possible to study the type of enhancement of a given area (Progressive/ Plateau/ Wash out).

Angiomammography has several advantages over breast MRI in the follow-up of chemotherapy: shorter examination time, shorter appointment time, better tolerated by the patients and without injection of Gadolinium chelates, which have recently been shown to cause definitive brain deposits during repeated injections. Currently, angiomammography is validated in the follow-up of breast cancers treated with neoadjuvant or primary chemotherapy, with an analysis of tumour response currently only morphological, as in breast MRI.

Here, the hypothesis is that the study of tumour enhancement by angiomammography may constitute a new predictive element of histological response: indeed, the performance of an initial angiomammography before treatment (baseline) and then a second angiomammography performed early in relation to the start of chemotherapy, could allow early prediction of which patients will have a complete histological response at the time of the closing surgery. This prospective study is to compare the variation in tumour enhancement, assessed on each of the two examinations using dedicated X-ray consoles, to the final histological result after closure surgery: it is hoped that the relative variation in tumour enhancement would be greater in responding patients.

ELIGIBILITY:
Inclusion Criteria:

* With a histological diagnosis of stage II or III localised breast cancer, with an indication for first or neoadjuvant chemotherapy validated by the RCP: HER2+, Triple negative
* Affiliated or beneficiary of a social security scheme or similar
* Having signed an informed consent for participation in the study.

Exclusion Criteria:

* Patients considered to be at very high risk (BRCA 1 and 2 mutation, Li Fraumeni syndrome, Lynch syndrome, previous thoracic irradiation for lymphoma) and high genetic risk as determined by an oncogenetic consultation
* Pregnancy, breastfeeding
* Contraindication to the injection of iodinated contrast material: hypersensitivity to the active substance or to one of the excipients of the contrast material, renal insufficiency with glomerular filtration rate < 35ml/min
* Patients who do not master the French language
* Patient who is an adult protected by law, under curatorship or guardianship
* Patient who has participated in another research study with a current exclusion period

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The evolution of the relative tumor enhancement (RTEe) (%) between the baseline and early re-evaluation CESM | At baseline, 2 and 8 months
  Evolution of the relative tumor enhancement (RTEe) between the baseline and early re-evaluation CESM (4-6 weeks after the start of chemotherapy). That is, the percentage of post-chemo tumor enhancement - Percentage of pre-chemo tumor enhancement / pre-chemo tumor enhancement
  The relative tumor enhancement (RTE) will be calculated as follows on each CESM (baseline and early follow up):
  RTE = (ROI 1 - ROI 2) / ROI 2
  The evolution of relative tumor enhancement (RTEe) between the initial CESM (RTEi) and the early follow-up CESM (RTEf) will be calculated.
  RTEe = (RTEf) - (RTEi) / (RTEi)

SECONDARY OUTCOMES:
RTEe according to the 3 categories of RCB score | At 8 months
  Evolution of the relative tumor enhancement (RTEe) according to:
  * RCB I: Minimal residual tumour
  * RCB II: Moderate response
  * RCB III: extensive residual tumour
The type of enhancement (TE) % | At baseline and 2 months
  The type of enhancement (%) will be calculated at each CESM (initial and follow-up) as follows :
  signal-to-noise ratio (SNR) on the late image - SNR on the early image / SNR on the late image.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France